CLINICAL TRIAL: NCT06363916
Title: Evaluation of Security and Efficacy of Medtrum Hybrid Closed Loop System in Children, Adolescents and Adults With Type 1 Diabetes
Brief Title: Evaluation of Security and Efficacy of Medtrum Hybrid Closed Loop System
Acronym: SEECLOOP
Status: Recruiting | Type: Observational
Sponsor: Medtrum France (Industry)
Collaborators: Axonal-Biostatem (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A00335-40
Record Dates: First submitted 2024-04-05; First posted 2024-04-12 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open Loop: Patients using the Insulin Management System device in a manual mode of operation. Patient must use the interface directly to deliver insulin. The algorithm will not be activated.
  Interventions: Device: Insulin Management System in Manual mode of operation
- Closed Loop: Patients using the Insulin Management System device in the Closed Loop mode of operation. The algorithm will be activated. The algorithm is capable of delivery of insulin based on sensor derived glucose levels, glucose level trends and insulin pump delivery history.
  Patients in this group can continue to an exploratory phase for the Automatic Meal Management function.
  Interventions: Device: Insulin Management System in Automatic mode of operation

INTERVENTIONS:
Device: Insulin Management System in Manual mode of operation — MEDTRUM A8 TouchCare® Insulin Management system which includes:
  * Patch pump: Pump base integrated with Hybrid Close Loop (HCL) algorithm not activated
  * Reservoir Patches
  * Continuous glucose monitoring (CGM): Glucose Sensor + Transmitter
  * Personal Diabetes Manager (PDM) and/or EasyPatch® App
  * EasyFollow® App, EasyView® website System is in conformity with EC marking n° HD 601 357 110001- TUV Rheinland dated February 19th of year 2019 and completed by system DoC 881160 dated June 30th of year 2020.
  EasyPatch mobile application is in conformity with EC marking n°709972 - BSI - dated March 6th 2020
  Groups: Open Loop
Device: Insulin Management System in Automatic mode of operation — MEDTRUM A8 TouchCare® Insulin Management system which includes:
  * Patch pump: Pump base integrated with Hybrid Close Loop (HCL) algorithm activated
  * Reservoir Patches
  * Continuous glucose monitoring (CGM): Glucose Sensor + Transmitter
  * Personal Diabetes Manager (PDM) and/or EasyPatch® App
  * EasyFollow® App, EasyView® website System is in conformity with EC marking n° HD 601 357 110001- TUV Rheinland dated February 19th of year 2019 and completed by system DoC 881160 dated June 30th of year 2020.
  EasyPatch mobile application is in conformity with EC marking n°709972 - BSI - dated March 6th 2020
  Groups: Closed Loop

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the MEDTRUM Hybrid Closed Loop (HCL) System in children, adolescents, and adults with type 1 diabetes (7-75 years old) in a home setting and to test the function of meal announcement in an extend study.

The main question it aims to answer is :

• Is the Hybrid Closed Loop system superior at increasing the time spent in the target glucose range of 70-180 mg/dL when compared to the Open (manual) Loop system ?

Participants will be :

* Trained into the use of the Insulin pump MEDTRUM A8 TouchCare® Insulin Management system
* Randomized to the Open Loop or Closed Loop group
* Respond to self administered questionnaires : the Hypoglycaemia Fear Survey, the Diabetes Quality of Life Questionnaire, and the Diabetes treatment Satisfaction Questionnaire status

Researchers will compare the time spent in the target glucose range of 70-180 mg/mL during the last 12 weeks of the study between the patients randomised to the Open Loop group and those randomised to the Closed Loop group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients living with Type 1 diabetes:

   * adults aged 18 to 75 years old (included)
   * children/adolescents aged 7 or older
2. Total daily dose of insulin ≥ 10 units per day & weighing >22 Kg
3. Patient and their parent(s)/guardian(s) trained and able to count carb
4. Current or previous insulin pump user or patient treated with multiple insulin injections
5. Patient glycaemic target is not achieved or suboptimal according to international consensus: HbA1c level equal and greater than 7% and less than 12% at the time of enrolment, or TIR < 70%, or TBR >4%
6. Any type of rapid insulin with a total daily insulin in the range of 10-60 IU (unauthorized use of insulin supplements by pen injector): Humalog™, Lyumjev (insulin lispro injection), Novorapid (insulin aspart) or FIASP® (" faster insulin aspart ")
7. Subject and their parent(s)/guardian(s) able to receive and understand study information, give written informed consent, and easily participate to the trial
8. Subject and their parent(s)/guardian(s) affiliated to the French social security system
9. Subject and their parent(s)/guardian(s) have the cognitive ability and can successfully operate all study devices and can adhere to the protocol

Exclusion Criteria:

1. Patient unable to tolerate tape adhesive, catheter or had any unresolved adverse skin condition and intolerance to steel
2. Patient not willing to perform finger stick blood glucose measurements required by the system and/or routine diabetes management
3. Patient with behaviour/lifestyle not compatible with optimal management of insulin therapy or deemed to be at significant risk of severe events (e.g. severe hypoglycaemia, diabetic ketoacidosis)
4. Unstable diabetic retinopathy
5. Pregnant women or planning to become pregnant during the study or breast-feeding
6. Patient abusing alcohol
7. Patient using DPP-4 inhibitor, GLP-1 agonists, metformin, or SGLT2 inhibitors during the last 3 months prior screening
8. Patient already participating in another interventional study
9. Patient currently using a hybrid closed loop system or patient who has stopped usage of Hybrid Closed loop system for less than 3 months
10. Patient under the protection of justice or under guardianship or curatorship, or hospitalised under duress or admitted to a health or social care establishment for purposes other than those of this investigation.

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 1 diabetes subjects with insulin therapy delivered by pump (aged over 7 years), current or previous insulin pump user or patient treated with multiple insulin injections.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Superiority of the algorithm on Time In Range (TIR) between the 2 randomised groups | V5 (6 months)
  Comparison between the 2 groups of the proportion of time spent in the target glucose range of 70-180 mg/dL based on sensor measured glucose concentrations during last 12 weeks of the study

SECONDARY OUTCOMES:
Evolution of TIR | V1 (Inclusion), V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months)
  Evolution of the time spent in the target glucose range of 70-180 mg/dL based on sensor measured glucose concentrations between visits V1-V2, V2-V4, V2-V5, in each group
Evolution of coefficient of glycemic variation | V1 (Inclusion), V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months)
  Evolution of coefficient of glycemic variation (CV) between visits V1-V2, V2-V4, V2-V5, and over the last 12 weeks period of the study, in each group
Superiority in Glycated Haemoglobin (HbA1c) improvement | V2 (Randomisation), V5 (6 months)
  Comparison between the 2 groups of the HbA1c change between visits V2 and V5
Evolution of Time spent Above Range (TAR) | V1 (Inclusion), V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months)
  Evolution of the time spent >180 mg/dL and >250 mg/dL, between visits V1-V2, V2-V4, V2-V5, and over the last 12 weeks period of the study, in each group
Evolution of Time spent Below Range (TBR) | V1 (Inclusion), V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months)
  Evolution of the time spent <54 mg/dL and <70 mg/dL, between visits V1-V2, V2-V4, V2-V5, and over the last 12 weeks period of the study, in each group
Body Mass Index change | V1 (Inclusion), V2 (Randomisation), V5 (6 months)
  Body Mass Index change (Mean value, Standard Deviation) between visits V1-V2, and V2-V5, in each group
Glucose sensor measurement change | V1 (Inclusion), V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months)
  Evolution of glucose sensor measurements (Mean value, Standard Deviation) between visits V1-V2, V2-V4, V2-V5, and over the last 12 weeks period of the study, in each group
Percentage of patients with TIR > 70% | V1 (Inclusion), V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months)
  Percentage of patients having spent >70% of their time in the target glucose range (70-180 mg/dL) between visits V1-V2, V2-V4, V2-V5, and over the last 12 weeks period of the study, in each group
Percentage of patients with TIR > 70% and TBR < 4%, and with TIR > 70% and TBR < 1% | V1 (Inclusion), V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months)
  Percentage of patients having spent >70% of their time in the target glucose range (70-180 mg/dL) and <4% of their time below range (54 to 70 mg/dL) and percentage of patients having spent >70% of their time in the target glucose range (70-180 mg/dL) and <1% of their time below range (54 to 70 mg/dL) between visits V1-V2, V2-V4, V2-V5, and over the last 12 weeks period of the study, in each group
Evolution of glucose management indicator (GMI) | V1 (Inclusion), V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months)
  Evolution of glucose management indicator values between visits V1-V2, V2-V4, V2-V5, and over the last 12 weeks period of the study, in each group
Evolution of dosage of insulin | V1 (Inclusion), V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months)
  Modification of total daily dose of insulin, of basal dose of insulin and bolus dose of insulin between Visit V1-V2, between visits V1-V2, V2-V4, V2-V5, and over the last 12 weeks period of the study, in each group
Time of device usage and time in automatic mode of insulin delivery (hybrid closed loop) | V1 (Inclusion), V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months)
  Time of sensor usage in percentage and time spent in Auto Mode during study
Evolution of Self-administered Questionnaires scores | V1 (Inclusion), V5 (6 months)
  Evolution of Self-administered Questionnaire Hypoglycaemia Fear Survey (HFS) score between visits V1 and V5
Evolution of Diabetes Treatment Satisfaction score | V1 (Inclusion), V5 (6 months)
  Evolution of Diabetes Treatment Satisfaction Questionnaire status (DTSQs) score between visits V1 and V5
Safety Events | V1 (Inclusion), V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months)
  Occurrence of Safety Events as defined by ISO 14155, including severe hypoglycaemia and ketoacidosis, local tolerance events related to devices (pump and sensor), incidents occuring with Medtrum devices

OTHER OUTCOMES:
Extension phase: Assessment of Automatic Meal Management function in Hybrid Closed Loop group on TIR | V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months), V6 (7 months)
  Evolution of the time spent in the target glucose range of 70-180 mg/dL based on sensor measured glucose concentrations between visits V2-V6 and V5-V6
Extension phase: Assessment of Automatic Meal Management function in Hybrid Closed Loop group on glucose sensor measurements | V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months), V6 (7 months)
  Evolution of glucose sensor measurements (Mean value, Standard Deviation) between visits V2-V6 and V5-V6
Extension phase: Assessment of Automatic Meal Management function in Hybrid Closed Loop group on TAR | V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months), V6 (7 months)
  Evolution of the time spent >180 mg/dL and >250 mg/dL, from V2 to V6, and V5 to V6
Extension phase: Assessment of Automatic Meal Management function in Hybrid Closed Loop group on TBR | V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months), V6 (7 months)
  Evolution of the time spent <54 mg/dL and <70 mg/dL, from V2 to V6, and V5 to V6
Extension phase: Assessment of Automatic Meal Management function in Hybrid Closed Loop group on GMI | V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months), V6 (7 months)
  Evolution of glucose management indicator values from V2 to V6, from V5 to V6
Extension phase: Assessment of Automatic Meal Management function in Hybrid Closed Loop group on dosage of insulin | V2 (Randomisation), V3 (1 month), V4 (3 months), V5 (6 months), V6 (7 months)
  Modification of total daily dose of insulin, of basal dose of insulin and bolus dose of insulin from V2 to V6, from V5 to V6
Extension phase: Assessment of Automatic Meal Management function in Hybrid Closed Loop group on Self-administered Questionnaires scores | V5 (6 months), V6 (7 months)
  Evolution of Diabetes Treatment Satisfaction Questionnaire status (DTSQs) score between visits V5 and V6

CONTACTS AND LOCATIONS:
Overall Officials: Freddy PENFORNIS, Principal Investigator — Centre Hospitalier Sud-Francilien, Corbeil
Locations (17):
- France (17):
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU Caen, Caen
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - Centre Hospitalier de Gonesse, Gonesse
  - Centre Hospitalier Saint-Louis, La Rochelle
  - Hôpital Hôtel-Dieu, Le Creusot
  - Hospices Civils de Lyon, Lyon
  - Hôpital Européen, Marseille
  - Hôpital La Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Hôpital Lariboisière, Paris
  - Hôpital Necker, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided